CLINICAL TRIAL: NCT05779384
Title: Frequency and Predictors of Exacerbations Within a COPD Population in Uganda
Brief Title: The COPD Attack Study
Acronym: COPA
Status: Completed | Type: Observational
Sponsor: Makerere University (Other)
Collaborators: GlaxoSmithKline (Industry); University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: MHREC1541
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Exacerbation COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: It was an observational study — data collected concerning the incidence of exacerbations

SUMMARY:
The goal of this observational study is to evaluate the frequency and predictors of exacerbations in COPD patient population in Uganda.

The main questions it aims to answer are:-

1. What is the proportion of frequent exacerbators (≥2/year) and what factors are associated with the frequent exacerbator phenotype?
2. What is the frequency of exacerbations and what factors are correlated with exacerbation frequency? Participants will be asked to offer demographic ,clinical and exposure questions. Questionnaires assessing disease burden, and quality of life will be administered. Clinical measurements, and complete blood count will be collected ta baseline and on sick visits. Spirometry will be measured at baseline and on the last visit. Samples will be collected for storage. Participants will be followed up for one year.

DETAILED DESCRIPTION:
In this prospective observational study aimed at evaluating the frequency and predictors of exacerbations in a COPD population, the following were the objectives.

Primary objective

1. To estimate the proportion and predictors of frequent COPD exacerbations in Ugandans with COPD. Secondary objective(s)

1. To determine the frequency and predictors of exacerbations among COPD patients in Uganda
2. To evaluate the aetiologies of COPD exacerbations including eosinophilia, and bacterial causes.
3. To evaluate outcomes such as quality of life, lung function decline in patients with exacerbations by frequency of the exacerbations. COPD will be diagnosed as follows Definitions and diagnostic criteria for COPD and its grading, and that of an exacerbation have been provided by the GOLD guidelines 4 . This study will use the GOLD definitions and classifications. As per GOLD 2018 guidelines 4 , COPD will be considered in any patient with appropriate spirometry who has dyspnea, chronic cough or sputum production, and/or a history of exposure to risk factors for the disease.

GOLD 2018 definition of an exacerbation:

An acute worsening in respiratory symptoms that results in additional therapy. A) Mild exacerbation: Requires additional treatment with short acting bronchodilators only B) Moderate exacerbation: Requires additional treatment with short acting bronchodilators plus antibiotics and / or oral corticosteroids C) Severe exacerbation: Requires hospitalization or visit to emergency room. participants will be followed up at three monthly intervals, except when they have had a severe exacerbation, where they will be followed up at two weekly intervals until they stabilise.

During the follow up visit, participant's COPD diaries will be evaluated for exacerbation length, severity and frequency as well as health care utilization. Additionally the CAT, CCQ and MRC dyspnoea scale questionaires, to evaluate the impact of COPD on quality of life will be administered. Finally lung function will be evaluated by spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥30yrs
* COPD diagnosis as per protocol (page 7)
* Attending URAC clinic sites
* Written informed consent
* Able to fill in diary or has attendant who can help fill it out
* Willing to attend follow up visits as required by study

Exclusion Criteria:

* Active pulmonary tuberculosis
* Other important co-morbid disease likely to affect participation or outcomes, such as lung cancer, asthma and any other that may be deemed so, in which case be discussed on case by case basis by the investigational team.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit COPD patients aged ≥ 30, diagnosed as specified on page 7. These patients will be identified during the screening phase as having GOLD airflow obstruction severity grades 1-4 and symptom/exacerbation risk categories A-D per the GOLD 2018 criteria (Figure 1). The cut-off of 30 years was chosen because prevalence studies in Ugandans indicated that COPD was prevalent in those as young as 30 years 18 .
Sampling Method: Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion and predictors of frequent exacerbators in a COPD patient population in Uganda | 1 year period of follow up
  The proportion of participants who had more than 2 exacerbations in the period of follow up and factors associated with these

SECONDARY OUTCOMES:
Frequency and predictors of exacerbations (e.g infections, biomarkers) in this patient populations | one year
  The frequency of exacerbations that participants developed and the factors associated with these

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Alupo, MMED, Principal Investigator — alupopat@gmail.com
Locations (2):
- Uganda (2):
  - Makerere University college of health sciences, Mulago National Referal Hospital Complex, Kampala
  - Makerere University Lung Institute, Kampala